CLINICAL TRIAL: NCT02487719
Title: Effektivität Der in Der Schwangerschaftsvorsorge routinemässig Angewandten Eisenprophylaxe
Brief Title: Different Iron Supplements for Prevention of Anemia in Pregnancy
Acronym: EDISA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0475
Record Dates: First submitted 2015-06-09; First posted 2015-07-01 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Iron-Deficiency Anemia; Pregnancy
Keywords: Iron deficiecy; pregnancy; prenatal care
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Iron-Dextran Complex; teferrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Iron sulfate (Active Comparator): Iron sulfate (or) is given if randomly asigned in this group and Ferritin at inclusion < 50 mcg/L.
  intervention: oral iron sulfate 1 tbl daily until birth
  Interventions: Drug: Iron sulfate and Iron polymaltose for prevention of iron deficiency anemia
- Iron polymaltose (Active Comparator): Iron polymaltose (or) is given if randomly asigned in this group and Ferritin at inclusion < 50 mcg/L.
  intervention: oral iron polymaltose 1 tbl daily until birth
  Interventions: Drug: Iron sulfate and Iron polymaltose for prevention of iron deficiency anemia
- Multimineral (No Intervention): Routine supplementation of multivitamin. multimineral only. Ferritin level > 50 mcg/L at inclusion. No additional iron supplementation.
  oral multivitamin- multimineral preparation 1 tbl daily until birth as done in daily clinic routine

INTERVENTIONS:
Drug: Iron sulfate and Iron polymaltose for prevention of iron deficiency anemia
  Other Names: gynotardiferon; maltofer; elevit
  Arms: Iron polymaltose; Iron sulfate

SUMMARY:
Examination of iron supplements routinely used in pregnancy to compare these with one another regarding effectiveness in the prevention of iron deficiency.

Determination of ferritin / hemoglobin every pregnant woman under the first routine check. Classification into one of three subgroups (group 1: iron sulfate, Group 2: iron polymaltose, Group 3: multivitamin- multimineral) depending on the measured values. Repetition of hemoglobin every 8 weeks, at the entrance to birth and postpartum day 1, additional provision of ferritin at the entrance to birth. In addition, registration of each child's birth weight and gestational age.

DETAILED DESCRIPTION:
Worldwide, iron deficiency is the most common shortage in women of childbearing age and also the most common cause of anemia. The prevalence of iron deficiency in young not pregnant women is 10-30%. During pregnancy take Frequency and importance of iron deficiency. Through organic growth and development of fetoplacental Unit and by maternal tissue formation, uterus growth and strong Expansion of maternal blood volume increases the pregnant woman the iron requirement for a Multiple. Starting from a non-pregnant state in the daily requirement of about 1 mg increasing this to 4-5 mg. Even with optimum food selection and a secured Increase of intestinal absorption in pregnancy, there is a negative Iron balance. The consequences are a depletion of iron stores (Serum ferritin <15 mcg / L) and a qualitative and quantitative disturbance of maternal Erythropoiesis with increased hypochromic and microcytic erythrocytes up to the occurrence anemia. The increased iron requirement is the background to a general recommendation an iron prophylaxis during pregnancy. However, this is possible due Reinforcement of gastrointestinal symptoms usually only from the 12th week of pregnancy is recommended. All pregnant women receive from the 12th week of pregnancy a multivitamin supplementation for the most important trace elements and vitamins. According to the guidelines of the Department of Obstetrics of USZ should a pregnant woman after the 12th week of pregnancy at a marginal ferritin <50mcg / l prophylactically receive additional iron and so anemia can be prevented. The aim of the study is on the one hand today's conventional iron supplements Maltofer Fol and Gyno-Tardyferon to examine their effectiveness, in particular with regard to the difference between two- and trivalent iron. On the other hand are at the usual multivitamin supplements. Women with normal iron stores at the beginning with respect to their effectiveness in preventing a depletion of these stores will be examined. Another aspect to be examined the occurrence of manifest iron deficiency anemia among called iron prophylaxis.

According to ferrtin value at first pregancy check, patients are enrolled after informed consent.

ferritin >50 mcg/L means patient will be randomized in eiter iron sulfate or iron polymaltose group. Ferritin > 50 mcg/L means pt will reeive multivitamin - multimineral containing iron. At midpregancy ferritin value is routinely checked as well at entering delivery floor at term.

ELIGIBILITY:
Inclusion Criteria:

* age above 18 yrs, singelton rpegnancy, inclusion before 16 completed weeks of gestation

Exclusion Criteria:

* multiple pregnancy, contraindication for oral iron supplements or mulltivitamin preparations
* iron deficiency or other anemia
* hemoglobinopatheis
* clinically significant disorders, as renal insuffisciency, hepatic dysfunction, cardiovascular disease

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-06 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin before delivery | up to 32 weeks
  anemia prevalence at delivery

SECONDARY OUTCOMES:
Birthweight | measured once at birth
  birthweight at term
Gestatonal age at birth | measured once at birth
  percentage of preterm delivies in each arm
Discontinuation of iron or mulimineral supplementation | delivery
  discontinuation rate in every arm
Ferritin before delivery | up to 32 weeks
  body iron stores at delivery

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Krafft, MD, Principal Investigator — University Hospital Zurich, Div. of Obstetrics
Locations (1):
- University Hospital Zurich, Dept of Obstetrics, Zurich, Canton of Zurich, Switzerland